CLINICAL TRIAL: NCT07370324
Title: From Knowledge to Confidence: The Effect of a Stoma Educational Program on Self-Care Practices and Life Satisfaction of Urostomy Patients
Brief Title: Stoma Educational Program on Self-Care Practices
Acronym: 0841
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Abubakr Mohamed Salama, Assist prof, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Stoma Educational Program
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Urostomy Patients; Self-Care Practices
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): routine hospital care
- study group (Experimental): receive educational intervention
  Interventions: Other: education

INTERVENTIONS:
Other: education — Educational intervention will be implemented to urostomy patients in multiple sessions, which will be divided into theoretical and practical sessions as following:
  Theoretical session:
  This part will include knowledge about anatomy and physiology of urinary system, pre and post operative care, complication and life style modifications…etc.
  Practical session:
  This session will cover care of urostomy including pouch system, changing of pouch, empty of pouch, self- catheterization and irrigation of urostomy.
  Arms: study group

SUMMARY:
provide a stoma educational program and evaluate the self-care practices and life satisfaction of urostomy patients.

DETAILED DESCRIPTION:
The data will be collected from urostomy patients and their medical records to establish a baseline for their knowledge and educational needs. The researcher will provide an illustrated colored instructional booklet. designed educational intervention will be implemented on urostomy patients in multiple sessions

ELIGIBILITY:
Inclusion Criteria:

* can communicate verbally
* accepted to engage in the study

Exclusion Criteria:

* psychiatric patients
* patient with chronic diseases that interfere with their self-care activities as

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
knowledge mean score | Evaluation of patients' knowledge immediately post and 3 months later
  measured by a questionnaire designed in the form of multiple-choice questions. Each answer receives one degree, with the exception of unknown and missed answers, which receive zero points. The scores obtained for each question were summed up to get the total score for the patients' knowledge.
Self-care mean score | Evaluation of patients' knowledge immediately and 3 months later
  Standardized, numerical, validated, and evidence-based measures are used to assess the stoma self-care abilities of patients undergoing UD. It comprises seven skills required to change a urostomy pouch system. Each ability was graded on a four-point scale, with values ranging from 0 to 3.
Self-efficacy mean score | Evaluation of patient self- efficacy immediately post- operative and 3 months later
  It is designed to assess a general sense of perceived self-efficacy, aiming to predict how individuals cope with daily hassles and adapt after experiencing various stressful life events, in addition to the challenges posed by the disease. Patients' responses will be categorized as follows: 1 = not being confident at all, 2 = slightly confident, 3 = fairly confident, 4 = highly confident, and 5 = extremely confident. High scores refer to positive self-efficacy, i.e., the subjective presence of ability. So the total score is 100, whereas less than 50 = low (-ve) self-efficacy and more than 50 = high (+ve) self-efficacy.

SECONDARY OUTCOMES:
quality-of-life mean score | Assess patients' quality of life 3 months later
  The urinary diversion quality of life questionnaire designed to assess quality of life for urinary diversion patients. It consists of questions that explored general condition and physical condition, reconstruction-related symptoms, psychological status, sexual life, social status, and satisfaction with the treatment. Patients' responses were categorized as follows: 1- not at all, 2- a little, 3- much, 4- very much.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Al Mansurah, Egypt